CLINICAL TRIAL: NCT07132866
Title: Prevention of Alcohol Use and Promotion of Well-being Among Middle School Students: A Randomized Controlled Trial of ADAPT
Brief Title: Randomized Controlled Trial of ADAPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADAPT_160172; ID: 160172 (Other Grant/Funding Number: TrygFonden, Denmark); ID: BSS-2025-056-S2 (Registry Identifier: Research Ethics Comittee, Aarhus University, Denmark)
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Prevention intervention; Neurodevelopmentally informed; Adolescents; Middle school; Alcohol; Parents; Prosocial

STUDY DESIGN:
Intervention Model Description: The study employs a 2-condition cluster randomized controlled trial design with two conditions: 1) ADAPT intervention, 2) Delayed Treatment (ADAPT intervention offered after the last follow-up)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT (Experimental): The ADAPT condition consist of the ADAPT intervention (group sessions with students, meeting with parents).
  Interventions: Behavioral: ADAPT
- Delayed Treatment Condition (DTC) (No Intervention): The control condition is a DTC. All adolescents in the DTC will receive assessments on the same timeline as ADAPT adolescents, but will not receive the intervention. Following the final 3-months follow-up survey, ADAPT will be offered to DTC students and their parents.

INTERVENTIONS:
Behavioral: ADAPT — The ADAPT intervention consists of three group sessions (of 75-90 min), with 6-8 8th grade students in each group, administered over three consecutive weeks, plus one interactive parent component (of 45 min) administered during the three weeks (separate from the student sessions).
  Arms: ADAPT

SUMMARY:
This trial examines the effectiveness of a novel neurodevelopmentally informed intervention - Adolescent Developmentally-Appropriate health Promotion Therapy (ADAPT) - on preventing alcohol use and promoting well-being among students in middle school in a heavy adolescent alcohol use region (Denmark). Using a 2-condition cluster-randomized controlled trial of students in 8th grade (ages 13-15), the following hypotheses are tested:

1. Compared to adolescents in the Delayed Treatment Condition (DTC), ADAPT adolescents will show significant reductions in intentions to drink (primary outcome) from baseline to 3 months post intervention.
2. Compared to adolescents in the DTC, ADAPT adolescents will show significant reductions in alcohol use and alcohol-related consequences, and significant increases in well-being and life satisfaction (secondary outcomes) from baseline to 3 months.

Additionally, acceptability and feasibility is examined.

DETAILED DESCRIPTION:
The main aim of this trial is to examine the effectiveness of a novel neurodevelopmentally informed intervention - Adolescent Developmentally-Appropriate health Promotion Therapy (ADAPT) - on preventing alcohol use and promoting well-being among students in middle school in a heavy adolescent alcohol use region (Denmark). Furthermore, we aim to examine ADAPT's feasibility and acceptability with students in middle school, their parents, and with staff (e.g., teachers and principals), to inform and guide next step, larger scale randomized controlled trials.

The study employs a 2-condition cluster-randomized controlled design in 8th grade students (ages 13-15), with the following conditions:

1. ADAPT: ADAPT intervention (consisting of three group sessions with students and one meeting with parents per school class) will be conducted by study staff immediately after baseline.
2. Delayed Treatment: ADAPT is offered to interested schools after the 3-month follow-up survey is completed.

The following hypotheses are tested:

1. Compared to adolescents in the DTC, ADAPT adolescents will show significant reductions in intentions to drink (primary outcome) from baseline to 3 months post intervention.
2. Compared to adolescents in the DTC, ADAPT adolescents will show significant reductions in alcohol use and alcohol-related consequences, and significant increases in well-being and life satisfaction (secondary outcomes) from baseline to 3 months.

All participants will complete an online baseline survey pre-intervention and online follow-ups at 1- and 3-months. Due to the large target N (N=1000), we will randomize students (and schools) in two blocks. The primary and secondary outcomes will be analyzed using generalized estimation equations (GEE) to account for the nested data structure: repeated measures, nested within students, nested within groups, nested within school classes, nested within schools. Feasibility of ADAPT will be measured quantitatively via student enrollment and attendance in ADAPT groups sessions, and parent attendance in the parent meeting. Acceptability of ADAPT will be measured via surveys (students, parents) and interviews (school staff).

ELIGIBILITY:
Inclusion Criteria:

* Students starting 8th grade in August 2025 in one of the participating public middle schools
* Understand and speak Danish
* Able to give informed active consent with informed passive consent from parents/guardians

Exclusion Criteria:

- Not fulfilling inclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Intentions to drink | From baseline to 3 months post intervention
  Assessed by single items assessing intention to drink at least one unit of alcohol and intention to get drunk (dichotomized).

SECONDARY OUTCOMES:
Past month use of alcohol | From baseline to 3 months post intervention
  Assessed with single items on past month use.
Past month consequences of drinking | From baseline to 3 months post intervention
  Assessed by 14 items covering physical, social and mental issues related to hazardous use of alcohol, developed by the team for Danish adolescents based on previous Danish surveys and the Rutgers Alcohol Problems Index. Example items include blackouts, (emotional) hangovers, intimate contact that was later regretted, with yes/no response options (summed score).
Life satisfaction | From baseline to 3 months post intervention
  Assessed with the Brief Multidimensional Students' Life Satisfaction Scale (BMSLSS), which measures perceived life satisfaction across five life domains (family life, friends, school, self, and living conditions), with a 7-point scale ranging from 'terrible' to 'delighted'. The mean of the sum of the 5 items represents the total life satisfaction score.
Psychological well-being | From baseline to 3 months post intervention
  Assessed with the World Health Organization Five Well-being Index (WHO-5). The Index includes five positively phrased items, and participants rate how well each statement applies to them (past two weeks) using a 6-point scale, ranging from 'None of the time' to 'All of the time' (summed score: range 0-25) with a score of 25 representing the best possible quality of life).
Well-being in class | From baseline to 3 months post intervention
  Assessed by six items rated on a five-point scale from 'completely disagree' to 'completely agree' e.g., I feel accepted by the others in my class (summed score: range 0-30) with a score of 30 representing the best possible well-being in class.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine R Thomsen, PhD, Principal Investigator — Centre for Alcohol and Drug Research, Department of Psychology and Behavioral Sciences, Aarhus BSS, Aarhus University
Locations (1):
- Centre for Alcohol and Drug Research, Department of Psychology and Behavioral Sciences, Aarhus BSS, Aarhus University, Aarhus, Denmark, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
After the conclusion of the study, data from the study will be made available by the Centre for Alcohol and Drug Research, Aarhus University, upon reasonable request, and within the limitations set by the Danish data protection legislation and regulation.

REFERENCES:
- [Derived] Romer Thomsen K, Hareskov N, Caspersen CK, Lauenborg AM, Bergmann MG, Ornbol E, Wellnitz KB, Feldstein Ewing SW. Prevention of alcohol use and promotion of well-being among middle school students: a study protocol for a randomized controlled trial of ADAPT. BMC Public Health. 2025 Nov 7;25(1):3840. doi: 10.1186/s12889-025-25037-5. PMID 41204109